CLINICAL TRIAL: NCT05205434
Title: Efficacy of Synchronous and Asynchronous Telerehabilitation in COVID-19 Discharges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Abdurrahman Tanhan, Research Assistant, Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BitlisErenU2
Record Dates: First submitted 2022-01-19; First posted 2022-01-25 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Telerehabilitation
Keywords: COVID-19; Telerehabilitation; Exercise program; Breathing exercises
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Synchronous telerehabilitation program (Video conference) (Experimental): Participants will exercise program at home for an average of 30 minutes a day, 3 days a week, under the supervision of a physiotherapist via synchronized video conference. The program will continue for 8 weeks. The exercise program will consist of physical exercises (aerobic and strength exercises) along with breathing exercises and an educational program. Physical exercises will be adjusted in 3 different difficulty levels: sitting, standing with or without support.
  Interventions: Other: Synchronous telerehabilitation programme
- Asynchronous telerehabilitation programme (Mobil app.) (Experimental): The same exercises as in the synchronous telerehabilitation program will be done at the same frequency. Participants will watch the videos sent by the investigator via the mobile application and then do the exercises at home. The participants will meet with the investigator once a week to an update exercise program.
  Interventions: Other: Asynchronous telerehabilitation programme
- Control (No Intervention): Participants in this group will only receive an educational program

INTERVENTIONS:
Other: Synchronous telerehabilitation programme — Exercise program and educational program
  Other Names: Video conference
  Arms: Synchronous telerehabilitation program (Video conference)
Other: Asynchronous telerehabilitation programme — Exercise program educational program
  Other Names: Mobil application
  Arms: Asynchronous telerehabilitation programme (Mobil app.)

SUMMARY:
Investigators aimed to evaluate the effectiveness of exercise programs given by synchronous and asynchronous telerehabilitation methods in patients after discharge from COVID-19.

DETAILED DESCRIPTION:
Fifty seven participants will be enrolled. Participants will be randomly divided into 3 groups.

For this purpose, patients will be recruited at the time of discharge from the hospital and two experimental groups with the same physical therapy and educational program will be carried out. participants in the control group will only educational program. Participants in experimental groups will be followed using videoconference interviews from synchronous telerehabilitation methods and mobile application from asynchronous telerehabilitation methods at home. These participants will be given an 8-week exercise program. The exercise program will consist of physical exercises (aerobic and strength exercises) along with breathing exercises and the patients will be evaluated before and after the treatment.

After treatment programs, the functional capacity, performance, and hemodynamic parameters of the participants will be evaluated. Quality of life, physical activity level, anxiety-depression, and fatigue severity will also be evaluated with questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients in the subacute period discharged
* Be 18 years or older
* Having received oxygen therapy or mechanical ventilation support in the hospital
* Access to online interviews and web-based exercises with a secure internet connection
* Having sufficient speaking and hearing skills for telerehabilitation
* Volunteer to participate in research

Exclusion Criteria:

* Unstable clinical condition
* Having had cerebrovascular disease, intra-articular drug injection or surgery of the lower extremities in the last 6 months
* Inability to walk independently, even with an assistive device
* Having serious neuromuscular problems
* Not being cooperative enough to answer and understand questionnaires and scales

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-09-25 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Incremental Shuttle Walk Test (ISWT) | Change from baseline walking distance (meters) of the patients at the end of the 8th week and, postintervation sixth months
  The participant will be asked to walk around two 9-meter cones and complete them within the given time. Oxygen saturation and heart rate will be measured before and immediately after the test. They will be asked to self-report dyspnea and fatigue according to the modified Borg scale (0-10).

SECONDARY OUTCOMES:
30-Second Chair Stand Test (30 CST) | Change from baseline number of sitting and staying of the patients at the end of the 8th week and, postintervation sixth months
  The patient will be asked to sit and stand as much as possible within 30 seconds, with his hands crossed over his chest. The number of sitting and staying for 30 seconds will be noted.
Brief Physical Performance Battery (BPPB) | Change from baseline score of the patients at the end of the 8th week and, postintervation sixth months
  It is a test used to evaluate the lower extremity function of patients. This battery represents the sum of 3 functional tests such as standing stance tests, 4 meters walking test and 5 times chair sit and stand (5STS). Each test is scored between 0 (not completing the test) and 4 (highest performance level)

OTHER OUTCOMES:
Oxygen Saturation and Heart Rate | Change from baseline oxygen saturation (SaO2) and heart rate (beats per minute) of the patients at the end of the 8th week and, postintervation sixth months
  Participants' resting oxygen saturation and heart rate, and oxygen saturation and heart rate after the tests will be evaluated
Dyspnea and Fatigue Level | Change from baseline dyspnea and fatigue of the patients at the end of the 8th week and, postintervation sixth months
  Participants' dyspnea and fatigue level, and dyspnea and fatigue level after the tests will be evaluated according to the Modified Borg (0-10) scale
Timed Up-Go Test (TUG) | Change from baseline time (second) of the patients at the end of the 8th week and, postintervation sixth months
  Participants are asked to get up from the chair, walk 3 m at a comfortable and safe pace, return and sit back in the chair.
International Physical Activity Questionnaire Short Form (IPAQ) | Change from baseline metabolic equivalent (MET)-minute/week of the patients at the end of the 8th week and, postintervation sixth months
  It is a scale used to determine the level of physical activity in adults. The scale questions vigorous and moderate physical activity, walking time of at least 10 minutes and daily sitting time in the last 7 days.
Hospital Anxiety Depression (HAD) Scale | Change from baseline score in scale of the patients at the end of the 8th week and, postintervation sixth months
  The questionnaire, which was filled in by the patient and includes the anxiety and depression subscales, consists of 14 items. Responses are scored between 0-3.
Fatigue Severity Scale | Change from baseline score in scale of the patients at the end of the 8th week and, postintervation sixth months
  This scale is a 9-item scale that measures the severity of fatigue in patients and its effect on one's activities and lifestyle. Responses are scored on a seven-point scale with 1 = strongly disagree and 7 = strongly agree.
Quality of Life Scale: Short Form-36 (SF-36) | Change from baseline score in scale of the patients at the end of the 8th week and, postintervation sixth months
  The self-assessment scale consists of 36 items and 8 sub-dimensions. The scale is evaluated considering the last four weeks. On the scale, 0 points indicate poor health and 100 points indicate good health.

CONTACTS AND LOCATIONS:
Overall Officials: Abdurrahman TANHAN, MSc, Principal Investigator — Bitlis Eren University
Locations (1):
- Marmara University, Maltepe, Istanbul, Turkey (Türkiye)